CLINICAL TRIAL: NCT05065541
Title: A Phase 1, Open-label, Multi-part Positron Emission Tomography (PET) Imaging Study to Evaluate the Biodistribution and Radiation Dosimetry of the Monoacylglycerol Lipase (MGLL) PET Ligand [18F]T-401 and to Evaluate Fatty Acid Amide Hydrolase (FAAH) and MGLL Enzyme Availability in the Central Nervous System Using [11C]MK-3168 and [18F]T-401 PET Ligands Before and After Oral Administration of Single and Multiple Doses of CC-97489 in Healthy Adult Subjects
Brief Title: Positron Emission Tomography (PET) Imaging Study to Evaluate Enzyme Availability in the Central Nervous System Before and After CC-97489 Administration in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-97489-CP-002; 2021-000646-17 (EudraCT Number)
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteers
Keywords: CC-97489; Healthy Adults; Phase 1; Positron Emission Tomography (PET) Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental)
  Interventions: Drug: [18F]T-401
- Part 2 (Experimental)
  Interventions: Drug: CC-97489; Drug: [18F]T-401; Drug: [11C]MK-3168
- Part 3 (Experimental)
  Interventions: Drug: CC-97489; Drug: [18F]T-401

INTERVENTIONS:
Drug: CC-97489 — Specified dose on specified days
  Arms: Part 2; Part 3
Drug: [18F]T-401 — Specified dose on specified days
Drug: [11C]MK-3168 — Specified dose on specified days
  Arms: Part 2

SUMMARY:
The purpose of this study is to evaluate enzyme availability in the central nervous system before and after CC-97489 administration in healthy participants

ELIGIBILITY:
Inclusion Criteria:

* Has a Body Mass Index (BMI) of 18.0 to 33.0 kg/m^2, inclusive. BMI = weight (kg)/(height [m])^2
* Must be healthy based on medical history, physical examination (PE), clinical laboratory test results, vital signs, and 12-lead electrocardiogram (ECG) at screening and check-in

Exclusion Criteria:

* Has any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
* Is pregnant or breastfeeding
* Is part of the study site staff personnel or a family member of the study site staff

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Radiation dosimetry calculated from PET-CT images | 1 day
Calculated % Injected Dose in brain and other key organs and tissues | 1 day
Calculated Standard Uptake Volume in brain and other key organs and tissues | 1 day
Change from baseline in SUV in the brain based on PET scans | Up to 14 days
Change from baseline in VT in the brain based on PET scans. | Up to 14 days

SECONDARY OUTCOMES:
Incidence of AEs | Up to 28 days after the last dose
Incidence of serious adverse events (SAEs) | Up to 28 days after the last dose
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: PR interval | Day 21
  PR interval: The time from the onset of the P wave to the start of the QRS complex
Incidence of clinically significant changes in ECG parameters: QRS interval | Day 21
  QRS interval: A combination of the Q wave, R wave and S wave, the "QRS complex" represents ventricular depolarization.
Incidence of clinically significant changes in ECG parameters: QT interval | Day 21
  QT interval: Measured from the beginning of the QRS complex to the end of the T wave.
Incidence of clinically significant changes in ECG parameters: QTcF interval | Day 21
  QTcF interval: Corrected QT interval using Fridericia's formula (QTcF).
Incidence of clinically significant changes in vital signs: Body temperature | Day 21
Incidence of clinically significant changes in vital signs: Respiratory rate | Day 21
Incidence of clinically significant changes in vital signs: Blood pressure | Day 21
Incidence of clinically significant changes in vital signs: Heart rate | Day 21
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Up to Day 18
Incidence of clinically significant changes in clinical laboratory results: Clinical Chemistry tests | Up to Day 18
Incidence of clinically significant changes in clinical laboratory results: Urinalysis tests | Up to Day 18
Pharmacokinetics - Maximum observed plasma concentration (Cmax) | Up to 19 days
Pharmacokinetics - Time to maximum observed plasma concentration (Tmax) | Up to 19 days
Pharmacokinetics - Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-∞) | Up to 19 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 001, Leuven, Vlaams Brabant, Belgium

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html